CLINICAL TRIAL: NCT03743467
Title: Study Regarding the Realization of a Standardized Protocol for the Evaluation of the Visual Condition in Parkinson's Disease
Brief Title: Study on the Visual Condition in Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Nicola Modugno, Neurologist, Head of Parkinson Center, Neuromed IRCCS
Other Study IDs: NMOD_01
Record Dates: First submitted 2018-11-07; First posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; vision; quality of life
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Health subjects
  Interventions: Diagnostic Test: Clinical evaluation of vision and eye tests
- PD patients Hoehn Yahr 1: Patients with Hoehn Yahr stage 1
  Interventions: Diagnostic Test: Clinical evaluation of vision and eye tests
- PD patients Hoehn Yahr 2-3: Patients with Hoehn Yahr stage 2 and 3
  Interventions: Diagnostic Test: Clinical evaluation of vision and eye tests

INTERVENTIONS:
Diagnostic Test: Clinical evaluation of vision and eye tests — * VFQ-25 Questionnaire
  * BCVA
  * Contrast sensitivity
  * Color sensitivity examination (Ishihara test 38 plates)
  * Complete evaluation of orthoptic features, eye movements, eyelid function, pupil function
  * Slit lamp examination
  * Shirmer test, Break up time test
  * Corneal pachymetry (optical pachymetry)
  * IOP
  * Quantitative and qualitative analysis of the macular area and of the optical disc by OCT: RPE, RNFL and Neuroretine Layer

SUMMARY:
Non motor symptoms and signs in Parkinson's disease (PD) also include a series of visual deficits; deepening these aspects could be useful for a better management of symptoms, to standardize a specific protocol for the issues related to vision and also to understand how these aspects are important for the understanding of the mechanisms underlying the PD.

DETAILED DESCRIPTION:
In Parkinson's disease (PD) several non-motor signs and symptoms already occur in the early stages of the disease; the symptoms are diverse and these also involve visual difficulties which commonly affect the majority of patients and which gradually worsen the quality of life.

The most common malfunction produced by PD is the dysfunction of dopaminergic pathways that may be responsible for a series of visual deficits too:

* decreased visual acuity and decreased sensibility to light and color,
* strabismus and forms of sensory and eye movement dysfunctions,
* eyelid dysfunctions and dry eye syndrome

Moreover, in patients affected by PD, typical retinal features were discovered for the first time in 2004 by the use of OCT (Optical Coherence Tomography) such as:

* the reduction of the retinal nerve fiber layer (RNFL)
* a typical thinning of the macular thickness, even if with different results. In the follow-up of the PD, these retinal features, verifiable by the use of OCT, could be considered as a marker of the pathology.

For these reasons it may be useful:

* quantify in an objective manner how much the visual aspects affect the overall deterioration of the quality of life in patients with PD
* demonstrate the validity of a specific and integrated outpatient diagnostic protocol for the study of visual and ophthalmological disorders in patients with PD
* demonstrate the diagnostic role of early changes in macular thickness and of the optic disc in subjects suffering from PD using the OCT
* establish orthoptic evidence in patients with PD

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Patients affected by Parkinson's disease (PD) according to the diagnostic criteria of the United Kingdom Brain Bank, in the ON phase of their usual treatment
* Hoehn-Yahr Stage from 1 to 3
* Signature of the Informed Consent and of the privacy form

Exclusion Criteria:

* Patients with symptoms and signs compatible with atypical parkinsonism
* PD patients treated with antagonist drugs for central dopaminergic receptors (first and second generation antipsychotics) in the last 6 months before enrollment
* Patients suffering from other neurological diseases
* Patients with evident cognitive impairment (MMSE <24/30)
* Patients with manifest eye movement disorders prior to the diagnosis of PD.
* Patients with daltonism
* Patients with amblyopia
* Patients suffering from high anisometropia
* Patients suffering from advanced cataracts
* Patients suffering from glaucoma
* Patients suffering from maculopathy
* Patients suffering from pathologies of the optic nerve
* Patients with severe visual field deficits
* Patients with refractive defects above 5 diopters

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Patients affected by Parkinson's disease (PD) according to the diagnostic criteria of the United Kingdom Brain Bank, in the ON phase of their usual treatment (Hoehn-Yahr Stage from 1 to 3) coming from Parkinson's Center of Neuromed IRCCS Institute with signature of the Informed Consent and of the privacy form.
  2. Health subjects coming from Neurological Department of Neuromed IRCCS Institute with signature of the Informed Consent and of the privacy form.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-11-05 (Estimated); Primary Completion 2018-11-05 (Estimated); Study Completion 2019-05-26 (Estimated)

PRIMARY OUTCOMES:
Check the impact of visual condition on the quality of life in patients with PD through the use of questionnaires. | through study completion with an avarage of 6 months
  Quantify the impact of visual condition using the VFQ-25 (Visual Functional Questionnaire) in patients with PD through the main method of this questionnaire:
  all items are scored, each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points, respectively so that scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score. The lowest percentage is the better outcome for the visual condition.
Survey the validity of a specific diagnostic protocol for the evaluation of the visual condition in patients with PD. | through study completion with an avarage of 6 months
  Review the validity of a specific and integrated ambulatory diagnostic protocol for the study of visual and ophthalmological disorders through a visit protocol and exams designed specifically for patients with PD based on the evidence of visual conditions in the disease currently present in the scientific literature trough the best corrected visual acuity expressed in twentieths and the use of the SLOAN chart.
Survey the validity of a specific diagnostic protocol for the evaluation of the visual condition in patients with PD. | through study completion with an avarage of 6 months
  Review the validity of a specific and integrated ambulatory diagnostic protocol for the study of visual and ophthalmological disorders through a visit protocol and exams designed specifically for patients with PD based on the evidence of visual conditions in the disease currently present in the scientific literature trough the quantification of contrast sensitivity expressed by the CSC (contrast sensitivity curve) trough the use of the Contrast Sensitivity Chart 6 lines.
Survey the validity of a specific diagnostic protocol for the evaluation of the visual condition in patients with PD. | through study completion with an avarage of 6 months
  Review the validity of a specific and integrated ambulatory diagnostic protocol for the study of visual and ophthalmological disorders through a visit protocol and exams designed specifically for patients with PD based on the evidence of visual conditions in the disease currently present in the scientific literature trough the color sensitivity examination with the administration of the Ishihara test (38 plates) and results expressed by the Ishihara algorithm.
Survey the validity of a specific diagnostic protocol for the evaluation of the visual condition in patients with PD. | through study completion with an avarage of 6 months
  Review the validity of a specific and integrated ambulatory diagnostic protocol for the study of visual and ophthalmological disorders through a visit protocol and exams designed specifically for patients with PD based on the evidence of visual conditions in the disease currently present in the scientific literature trough the Shirmer test with results expressed in millimeters.
Survey the validity of a specific diagnostic protocol for the evaluation of the visual condition in patients with PD. | through study completion with an avarage of 6 months
  Review the validity of a specific and integrated ambulatory diagnostic protocol for the study of visual and ophthalmological disorders through a visit protocol and exams designed specifically for patients with PD based on the evidence of visual conditions in the disease currently present in the scientific literature trough the break up time test with results expressed in seconds of tear break.
Survey the validity of a specific diagnostic protocol for the evaluation of the visual condition in patients with PD. | through study completion with an avarage of 6 months
  Review the validity of a specific and integrated ambulatory diagnostic protocol for the study of visual and ophthalmological disorders through a visit protocol and exams designed specifically for patients with PD based on the evidence of visual conditions in the disease currently present in the scientific literature trough the measurement of ocular pressure expressed in mmHg by the use of a Non- Contact Tonometry.
Inspection of orthoptic condition in patients with PD | through study completion with an avarage of 6 months
  Analysis of orthoptic features in patients with PD trough eye movements examination to determine hypofunctions/ hyperfunctions in ductions and versions.
Inspection of orthoptic condition in patients with PD | through study completion with an avarage of 6 months
  Analysis of orthoptic features in patients with PD trough the quantification of convergence by the calculation of the near point of convergence expressed in millimeters.
Inspection of orthoptic condition in patients with PD | through study completion with an avarage of 6 months
  Analysis of orthoptic features in patients with PD trough the quantification of stereopsis expressed in seconds of arc trough the use of Lang stereo test and TNO stereo test.
Inspection of orthoptic condition in patients with PD | through study completion with an avarage of 6 months
  Analysis of orthoptic features in patients with PD by checking the presence of latent or manifest squint trough Cover and Uncover test in 9 position of gaze.
Inspection of orthoptic condition in patients with PD | through study completion with an avarage of 6 months
  Analysis of orthoptic features in patients with PD trough the quantification of the fusional amplitude expressed in prismatic diopters at distance (6 meters) and near (40 cm).
Observation of retinal features in patients with PD through the use of OCT | through study completion with an avarage of 6 months
  Registration of the retinal features in patients with PD using OCT trough a quantitative analysis of the macular area and of the optical disc by the registration of retinal tickness expressed in microns for RPE, RNFL and Neuroretine Layer.

CONTACTS AND LOCATIONS:
Overall Officials: Modugno Nicola, MD, PHD, Principal Investigator — Neuromed IRCCS
Locations (2):
- Italy (2):
  - Neuromed IRCCS, Pozzilli, Isernia
  - Irccs Neuromed, Pozzilli, Isernia